CLINICAL TRIAL: NCT00910338
Title: Efficacy and Safety of Extracorporeal Biofeedback Pelvic Floor Muscle Training to Treat Urodynamic Stress Incontinence
Brief Title: Efficacy and Safety of Extracorporeal Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KYU-SUNG LEE (Other)
Collaborators: Furun Medical (Industry)
Responsible Party: Sponsor-Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-06-075
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2011-04

CONDITIONS: Female Stress Urinary Incontinence
Keywords: Pelvic Floor Muscle Training; Extracorporeal Biofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PFMT with Extracorporeal Biobeedback (Experimental)
  Interventions: Device: PFMT with Extracorporeal Biofeedback

INTERVENTIONS:
Device: PFMT with Extracorporeal Biofeedback — Pelvic Floor Muscle Training with Extracorporeal Biofeedback Device for 12 weeks
  * Twice a week for the first 4 weeks
  * Once a week for the next 8 weeks
  Other Names: HnJ-5300

SUMMARY:
Stress urinary incontinence is the most common type of female incontinence. The efficacy of pelvic floor muscle training with biofeedback has been already proved in many studies. But intravaginal probe is one of the limitation. So, the purpose of this study is to assess the efficacy and safety of extracorporeal biofeedback device with pelvic floor muscle training.

ELIGIBILITY:
Inclusion Criteria:

* Women with stress urinary incontinence
* Standard pad test > 2gram

Exclusion Criteria:

Women with:

* Mixed urinary incontinence of which urgency incontinence is dominant
* True incontinence
* Overflow incontinence
* Treatment within 14 days preceding screening, or expected to initiate treatment during the study with electrostimulation, bladder training
* Treatment within 7 days preceding screening, or expected to initiate treatment during the study with OAB medication or other medication which affect bladder function
* Pelvic organ prolapse which the stage is at least 2
* Proven urinary tract infection during screening period
* Pacemaker
* Pregnant women
* Neurogenic voiding dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cure rate according to standard pad test ; Cure is defined as less than 2g on the standard pad test. | After 12 weeks of treatment

SECONDARY OUTCOMES:
Change in Incontinence severity VAS (I-VAS), Sandvik questionnaire, Incontinence Quality of Life (I-QoL), and Pelvic Floor Muscle Strength. | After 12 weeks of treatment
Patient perception of Treatment Benefit, Satisfaction, Willingness to Retreatment/Recommendation (BSW). | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Irwon-dong
  - Asan Medical Center, Ulsan College of Medicine, Seoul